CLINICAL TRIAL: NCT00623948
Title: Implanted Gluteal Stimulation System for Pressure Sore Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Suitable implanted technolgy was not available
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B4664-R
Record Dates: First submitted 2008-02-11; First posted 2008-02-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; Electrical Stimulation; Spinal Cord Injury
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Device: A fully implanted gluteal stimulation (GSTIM) system

INTERVENTIONS:
Device: A fully implanted gluteal stimulation (GSTIM) system — A fully implanted gluteal stimulation system

SUMMARY:
This project will evaluate the feasibility of using a fully implanted gluteal stimulation system for the prevention of Pressure ulcers. The specific goal of this study will be a pilot clinical trial of veterans with reduced mobility in order to establish clinical efficacy of a 2-channel bilateral gluteal stimulation system. A two-arm crossover study of wheelchair users with complete SCI will be carried out. All study participants will receive a fully implanted system incorporating implanted IM electrodes and a Micropulse I IPG stimulator (NDI Medical). Group assignments will be determined at enrollment using a modified randomization scheme. A total of 10 subjects will be recruited to the pilot clinical trial.

DETAILED DESCRIPTION:
Within the scope of the study the aims will be to: (1. Develop the pre-implantation assessment protocol utilizing targeted CT to locate optimal gluteal motor points bilaterally.) CT assessment of the pelvic region in spinal cord injured subjects will be carried out to determine regional vascular and nervous anatomy. This will allow us to achieve optimal electrode placement using a minimally invasive implantation procedure. (2. Develop the implanted gluteal stimulation system.) The fully implanted gluteal stimulation (GSTIM) system is envisioned as a marriage between the established technology of the implanted IM electrodes developed by the Cleveland FES Center and the newly developed Micropulse I 2-channel stimulator. The Micropulse I IPG is a small, rechargeable stimulator developed by NDI Medical as a platform technology for neuromodulation and neurostimulation applications. The device will be customized in order to provide two synchronized channels of stimulation for the GSTIM system. (3. Implement and evaluate implanted gluteal stimulation system in human volunteers.) A pilot clinical trial of the fully implanted gluteal stimulation system will be carried out using a two-arm crossover study of ten wheelchair users at risk for pressure ulcer development due to impaired mobility. Pre-defined selection criteria will be employed to screen potential participants physically and psychologically. All participants will receive a stimulation system consisting of implanted IM electrodes inserted bilaterally in the gluteus maximus together with the Micropulse I stimulator implanted subcutaneously in the lower abdomen. Tissue health will be assessed at three month intervals during the 12-month period following implantation. The clinical application of this system is of great relevance to the veteran population at risk of pressure ulcer development. The project will add value to the continued improvement in health care provision for veterans, allowing them to benefit from the most recent advances in medical device technology. Although the initial target user group is veterans with SCI, the proposes system will have applications to other patient populations at risk due to reduced mobility, such as those with multiple sclerosis and the elderly.

ELIGIBILITY:
Inclusion Criteria:

Motor and sensory complete SCI higher than the level T12.

Exclusion Criteria:

Eligible subjects will have had no open skin problems or hospitalizations during the three months prior to entrance into the study. Additional exclusion criteria relating to clinical factors and suitability include:

1. Age less than 18 years.
2. Less than two years post-injury or loss of independent walking ability.
3. More than three urinary tract infections in the previous year.
4. Significant active systemic disease, e.g. heart disease, renal failure, compromised renal function, diabetes.
5. Abnormal nutritional status based on albumin and total protein levels at recruitment (3.0 for albumin, 6.0 for total protein).
6. Osteomyelitis of the pelvic regional, indicated by positive pelvic inlet x-ray from routine annual urologic examination or bone scan.
7. Previous surgery in the perineal region that radically alters the basic anatomy, particularly regional innervation and blood supply., e.g., amputation, hemipelvectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcomes measures will be changes in tissue health variables and user satisfaction | baseline, 4 weeks, and six months

SECONDARY OUTCOMES:
Progressive changes in muscle bulk and tissue blood flow will be evaluated using CT scanning and transcutaneous oxygen measurement | baseline, 4 weeks, and six months
Pressure distribution changes over the long-term (due to muscle changes) and over the short-term (due to muscle contractions) will be assessed by interface pressure measurement. | baseline, 4 weeks, and six months

CONTACTS AND LOCATIONS:
Overall Officials: Kath M. Bogie, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States